CLINICAL TRIAL: NCT03755726
Title: A New Breath for Malignant Hypertension: Implementation of the HAMA Cohort
Acronym: HAMA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de PAU (Other)
Responsible Party: Principal Investigator, Romain Boulestreau, Principal Investigator, Centre Hospitalier de PAU
Other Study IDs: CHPAU2018/01
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Malignant Hypertension
MeSH Terms: conditions — Hypertension, Malignant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This registry aims to provide the first prospective, multicentric database of patients with malignant hypertension. It will allow to assess modern epidemiology of the disease, diversity of current management and care pathway, to deepen our pathophysiological knowledges, to modernize the definition of this form of hypertension and its diagnostic criteria. The network that will emerge will finally lead to the opportunity of setting up therapeutic trials and establishing recommendations based on solid scientific evidence.

DETAILED DESCRIPTION:
Malignant hypertension is the most severe form of high blood pressure, fatal if left untreated. It has not disappeared, with an increasing incidence. Patients with the disease, mainly young (35 to 55 years of age), have an unfavorable cardiovascular prognosis (14% of cardiovascular and renal events at 4 years). Despite these facts, scientific research on the subject remains limited. The definitions and diagnostic criteria have not changed since 1929, and the therapeutic recommendations remain empirical.

This first prospective and multicentric registry will increase and modernize the knowledge of the disease. From these data, diagnostic and therapeutic recommendations based on solid scientific evidence could be developed.

The investigators want to first recruit 500 patients and define their prognosis at 5 years. The impact of the patient's phenotype, type and number of target organs affected will be studied.

A modern definition, adapted to these results, could be proposed. The epidemiology of the disease, the care pathways, the target organ disorders and the management carried out in the centers will be described in detail.

ELIGIBILITY:
Inclusion Criteria:

* Malignant hypertension according to the classic definition (Severe hypertension, above 180/110 associated with severe hypertensive retinopathy)
* Severe hypertension (above 180/110) associated with acute damage of 3 target organ due to high blood pressure

Exclusion Criteria:

* Age < 18 years old
* Patients who cannot freely give their consent, or patients who refuse to participate
* Dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with malignant hypertension
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2019-09-20 (Actual); Primary Completion 2034-09-20 (Estimated); Study Completion 2034-09-20 (Estimated)

PRIMARY OUTCOMES:
prognosis | 5 years
  5-year prognosis for patients with malignant hypertension

CONTACTS AND LOCATIONS:
Locations (37):
- France (36):
  - CH d'Annecy, Annecy
  - CH de la côte Basque, Bayonne
  - Avicenne APHP, Bobigny
  - CHU - Hôpital St André, Bordeaux
  - CH de Chalon sur Saone, Chalon-sur-Saône
  - CH Métropole, Chambéry
  - CHU de Clermont FERRAND, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - CH de Dinard, Dinard
  - CHU Michallon, Grenoble
  - hôpital de Haguenau, Haguenau
  - Pôle Santé Sud, Le Mans
  - CH de Libourne, Libourne
  - CHRU de Lille, Lille
  - Clinique Vert Coteau, Marseille
  - Hopital de la conception, Marseille
  - CH Martigues, Martigues
  - CHU de Montellier, Montpellier
  - CHU - Hôpital Laennec, Nantes
  - Hôpital Saint Joseph, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - APHP Bichat, Paris
  - Fondation Adolphe de Rothschild, Paris
  - Hôpital Tenon, Paris
  - CH de PAU, Pau
  - CHU de Pointe à Pitre, Pitres
  - CHU de Poitiers, Poitiers
  - CHU de Rennes, Rennes
  - CHU de ROUEN, Rouen
  - Clinique sainte Clotilde, Saint-Denis
  - CHU de St Etienne, Saint-Etienne
  - CH de St Nazaire, Saint-Nazaire
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse Rangueil, Toulouse
  - CHU de Tours, Tours
  - CH de Valenciennes, Valenciennes
- National Institute of Cardiology, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boulestreau R, Lorthioir A, Dreau H, Persu A, Cremer A, Tharaux PL, Rubin S, Maier B, Mazighi M, Seris A, Paques M, Bonnin S, Halimi JM, Debeugny S, Gosse P; for the HAMA investigators. Baseline characteristics of the first 302 patients included for acute malignant hypertension crisis in the prospective multidisciplinary HAMA cohort. J Hypertens. 2024 Dec 1;42(12):2131-2138. doi: 10.1097/HJH.0000000000003851. Epub 2024 Oct 7. PMID 39351849